CLINICAL TRIAL: NCT06175195
Title: Psychoeducational Program for Treatment Refusal, Psychiatric Symptoms and Quality of Life Among Cancer Patients: A Randomized Control Trial
Brief Title: Psychoeducational Program for Cancer Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Government College University Faisalabad (Other)
Responsible Party: Principal Investigator, Qasir Abbas, Principal Investigator, Government College University Faisalabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GovernmentCUF
Record Dates: First submitted 2023-11-23; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Psychoeducation
Keywords: Psychoeducational Program.; Treatment refusal; Depressive symptoms; Anxiety; Help-seeking attitude; Cancer Patients
MeSH Terms: conditions — Treatment Refusal; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized control trial design would be used in this study. It would be two arm study and there would be two groups an experimental and wait-list control group. Experimental group will receive intervention and another group would be placed in waitlist. In this research, parallel group design would be used. We will give treatment to all participants in a parallel way. Allocation ratio and framework would be equivalence i.e., treatment group and control group would be equal number of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Experimental Group:
  Participants in the experimental group would receive 8-10 session of psychoeducational based Program.
  Waitlist control Group:
  Participants in the Control group would not receive psychoeducational Intervention.
  Interventions: Behavioral: Psychoeducational Inervention
- Control Group (No Intervention): Control Group:
  Participants in the control group did not receive the said psychoeducational intervention.

INTERVENTIONS:
Behavioral: Psychoeducational Inervention — Psychoeducational Program would be used as an intervention stratégie for cancer patients to provide understanding and insight to the patients about the problems. Further, this program would address treatment refusal and illness denial, depressive symptoms, and treatment related irrational fears and anxiety. Moreover, this program will improve patients' motivation and attitude toward changing health, and quality of life.
  Arms: Treatment Group

SUMMARY:
The main objective of the study are:

1. To explore the effectiveness of psychoeducation program for cancer patients who refuse treatment because of irrational fears and anxieties.
2. To explore the effectiveness of psychoeducation program for cancer patients who have negative attitudes, and low motivation toward treatment which causes depression and affects the quality of life.

DETAILED DESCRIPTION:
Participants:

In this Randomized control trial, N=200 participants would be enrolled for eligibility assessment from different cancer hospitals in Faisalabad and Lahore. 60 participants after the eligibility assessment and screening would be allocated to experimental and waitlist treatment conditions. Participants would be allocated through matchable group characteristics. In experimental group, the diagnosed patients of cancer who refuse psychotherapy would be included and 08 to 10 sessions of psychoeducation program would be provided. In waitlist treatment condition, diagnosed cancer patients would be taken. Each of the group will be comprised of n= 30.

Elegibility Criteria:

The participants that would be taken in the study would be diagnosed patients of cancer with stage I, II and III who refused psychological treatment as recommended by the practitioner. Second eligibility criteria of the participants would be at least mild score on PHD-9 to cross check the mental health problems. The patients would be taken from lower, middle and upper socioeconomic status and their age range would be from 20-70 years. The patients diagnosed with 4th stage would be excluded.

Interventions:

Psychoeducational Program would be used as an intervention stratégie for cancer patients to provide understanding and insight to the patients about the problems. Further, this program would address treatment refusal and illness denial, depressive symptoms, and treatment related irrational fears and anxiety. Moreover, this program will improve patients' motivation and attitude toward changing health, and quality of life.

Expected Outcomes This study would provide valuable information to the mental health practitioners to treat and develop the guidelines and protocol for patients with cancer. Psychoeducational Program played substantial role as supportive intervention to develop insight, motivation and positive attitude toward treatment as well as to enhance adherence to treatment among patients with cancer. And there would be substantial decrease in depression, treatment related fear and anxiety. Moreover, this program will improve patients' motivation and attitude toward changing health, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Participants who will be diagnosed with cancer at stage-I, II and III and who have refused medical and psychological treatment will be included in the treatment
* The second eligibility criterion of the participants would be at least mild score on PHD-9 to cross-check the mental health problems Participants they have diagnosed by the consultant after proper medical screening and evaluation will be included
* The patients would be taken from lower, middle and upper socioeconomic status.
* Their age range would be from 20-70 years.

Exclusion Criteria:

Participants with medical and psychiatric comorbidities will be excluded

• The patients diagnosed with 4th stage would be excluded. Participants with serious medical condition will be excluded

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-04-10 (Estimated)

PRIMARY OUTCOMES:
Treatment Refusal | 3-5 weeks
  Initially, we will enroll the patients for eligibility assessment and the eligible patients who are refusing medical (Chemotherapy, Radiation and Surgery) and psychological treatment (Counseling, psychotherapy) will be referred for psychological evaluations
Depression and Anxiety | after allocation (1 week)
  Depression will be assessed by using Patient Health Questionnaire-9. A Score of 5, 10, 15, and 20 correspond to categorizations of mild, moderate, moderately severe, and severe depression respectively. Hospital Anxiety and Depression will be assessed by using Hospital Anxiety and Depression Scale. A score of 0-7 is considered normal, 8-10 as borderline and 11-21 as either anxious or depressed
Illness denial | after allocation (1 week)
  Illness denial will be assessed by using Illness Denial Questionnaire. Higher score indicate high Illness denial whereas low score indicate low illness denial.
Motivation and Help-Seeking attitude | after allocation (1 week)
  Motivation will be assessed by using Motivation and attitude towards changing health Scale. Higher score indicate higher motivation whereas low score indicate low motivation.
  Mental Help seeking attitude will be assessed by using Mental Help Seeking Attitude Scale. Higher score indicate high mental help seeking attitude whereas low score indicate low mental help seeking attitude.
Quality of Life Scale | after allocation (1 week)
  Quality of Life will be measured by World Health Organization Quality of Life BREF. Higher score indicate high quality of life whereas low score indicate low quality of life

SECONDARY OUTCOMES:
Duration of illness | at the time of pre assessment (1 week)
  They will be assessed through interview information
stage of cancer | after allocation at pre-assessment (1 week)
  They will be assessed through history taking information

CONTACTS AND LOCATIONS:
Overall Officials: Qasir Abbas, PHD, Principal Investigator — Government College University, Faislabad.
Locations (1):
- Qasir Abbas, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No